CLINICAL TRIAL: NCT03307031
Title: The Influence of Pilates Exercises Training Volume on Metabolic, Physical Fitness and Quality of Life Outcomes in Dyslipidemic Women: A Controlled Clinical Trial.
Brief Title: The Influence of Pilates Exercises Training Volume on Metabolic Outcomes in Dyslipidemic Women.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Luiz Fernando Martins Kruel, Doctor, Federal University of Rio Grande do Sul
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1.990.955
Record Dates: First submitted 2017-09-13; First posted 2017-10-11 (Actual); Last update posted 2017-10-11 (Actual); Status verified 2017-08

CONDITIONS: Dyslipidemias
Keywords: training volume; elderly; lipid profile; postmenopausal
MeSH Terms: conditions — Dyslipidemias | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: A CONTROLLED CLINICAL TRIAL
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High Volume Group (Experimental): Performed four weekly sessions, during 10 weeks with 45 to 55 minutes per session.
  Interventions: Other: High Volume Group
- Low Volume Group (Experimental): Performed only twice a week, during 10 weeks with 45 to 55 minutes per session.
  Interventions: Other: Low Volume Group
- Control Group (Placebo Comparator): Did not exercise, during 10 weeks.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: High Volume Group — Performed four weekly session, during 10 weeks with 45 to 55 minutes per session.
  Arms: High Volume Group
Other: Low Volume Group — Performed only twice a week, during 10 weeks with 45 to 55 minutes per session.
  Arms: Low Volume Group
Other: Control Group — Did not exercise, during 10 weeks.
  Arms: Control Group

SUMMARY:
The aim of the present study was to assess the influence of different volumes of Pilates training exercises on metabolic, blood pressure (BP), functional physical fitness (PF) and quality of life (QL) outcomes in postmenopausal dyslipidemic women. In total, 26 women participated in the controlled clinical trial, being allocated into three groups: high volume group (HVG; n=9), low volume group (LVG; n=11) and control group (CG, n=6). HVG performed four weekly sessions and LVG performed only twice a week, during 10 weeks with 45 to 55 minutes per session. Before and after the intervention period, metabolic, BP, PF, QL and cardiovascular risk score (CRS) outcomes were measured. The results were described by mean values with lower and upper limits (95% confidence interval). Comparisons between groups and intra-groups were performed adopting Generalized Estimating Equations (GEE) method, with post hoc of Bonferroni and significance level of ɑ=0,05.

ELIGIBILITY:
Inclusion Criteria:

* Dyslipidemic, postmenopausal and sedentary.

Exclusion Criteria:

* Women taking statins and smokers.

Ages: 60 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-07-28 (Actual); Study Completion 2017-09-13 (Actual)

PRIMARY OUTCOMES:
Metabolic outcomes | 10 weeks
  Cholesterol (mg/dl)
Metabolic outcomes | 10 weeks
  Low-density lipoprotein (mg/dl)
Metabolic outcomes | 10 weeks
  Triglycerides (mg/dl)
Metabolic outcomes | 10 weeks
  High-density lipoprotein (mg/dl)
Metabolic outcomes | 10 weeks
  TC/HDL ratio

SECONDARY OUTCOMES:
Secondary outcomes | 10 weeks
  Systolic blood pressure (mmHg)
Secondary outcomes | 10 weeks
  Diastolic blood pressure (mmHg)
Secondary outcomes | 10 weeks
  Functional physical fitness
Secondary outcomes | 10 weeks
  Quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Adriana Cristine Koch Buttelli, Porto Alegre, Rio Grande do Sul, Brazil